CLINICAL TRIAL: NCT04250181
Title: HPvSP-AF Trail: Is High RF Energy Ablation of Atrial Fibrillation Fast, Safe, Less Painful and Effective - a Propensity Score Matched Analysis of 30/25W, 40W and 50W RF Energy Settings
Brief Title: High Power vs Standard Power RF Ablation of Atrial Fibrillation in Conscious Patients
Acronym: HPvSP-AF
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Maciej Wójcik, MD, PhD, Clinical Professor, Medical University of Lublin
Other Study IDs: HPvSP-AF ablation
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation ablation; high power radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard RF: ablation with RF power of 30 Watts (30W) and with 25 Watts (25W) on posterior wall
  Interventions: Other: RF ablation of atrial fibrillation
- High RF 40W (40 Watts): ablation with RF power of 40 watts (40W)
  Interventions: Other: RF ablation of atrial fibrillation
- High RF 50W (50 Watts): ablation with RF power of 50 watts (50W)
  Interventions: Other: RF ablation of atrial fibrillation

INTERVENTIONS:
Other: RF ablation of atrial fibrillation — Comparison of standard, 40W and 50W RF energy setting for ablation of atrial fibrillation

SUMMARY:
High RF energy ablation of atrial fibrillation is fast, safe, less painful and effective procedure.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) ablation is the most commonly performed radiofrequency (RF) ablation and is usually associated with a long procedural time and sensation of pain in conscious patients. Prolonged radiation exposure during the procedure puts the patient and the operator at risk of malignancy and genetic abnormalities. Complications such as asymptomatic cerebral lesions, tamponade, perforation, and also arrhythmia recurrence were associated with longer ablation time.

High-power, shorter-duration radiofrequency ablation (HPSDRFA) appears to be a novel concept for atrial fibrillation (AF) but there are scarce data in conscious patients. The lesion side index (LSI) value has been associated with durability of pulmonary vein isolation (PVI) lesions.

We hypothesised that HPSDRFA applications based on the lesion side index (LSI; its has been associated with durability of pulmonary vein isolation (PVI) lesions) which were not inferior to standard approach regarding safety and effectiveness with shorten procedure time and being less painful for a patient.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patients with non-valvular AF,
* aged:18-85, first procedure in left atrium,
* exclusion of thrombus in left atrium and left atrium appendage,
* left ventricle ejection fraction >55%

Exclusion Criteria:

* age below 18 or above 85 years,
* left ventricle ejection fraction<55%,
* previous procedure in left atrium,
* valvular AF

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-02-08 (Actual)

PRIMARY OUTCOMES:
Procedure time: | procedure
  Total procedure time (needle to needle time).

SECONDARY OUTCOMES:
Left atrial dwelling time | transeptal access to removal of a catheter and a sheath
  time of left atrium instrumentation
Voltage mapping time | procedure
  time needed to perform 3D electroanatomical map and high density voltage mapping of left atrium.
Total RF time | procedure
  time of all performed radiofrequency (RF) applications
Total number of RF applications | procedure
  number of all RF applications performed during a procedure
X-Ray time | procedure
  the total time of fluoroscopy
Complications | 12 months
  both procedure-related complications and all complications in 12 moths follow-up as follows: Cardiac tamponade/perforation [yes/no], Stroke/TIA (Transient ischemic attack) [yes/no], Oesophageal injury (perforation/fistula) [yes/no], Death (procedural related, one year follow up) [yes/no], Stem pops [yes/no], Catheter char [yes/no], Phrenic nerve paralysis [yes/no], PV stenosis requiring intervention [yes/no], Gastrointestinal bleeding or gastrointestinal complaints [yes/no], Need for periprocedural pacemaker implantation [yes/no], Vascular access complication which required intervention [yes/no], Vascular access complication which not required intervention [yes/no],
Number of stopped RF applications as a result of pain complained by a patient | procedure
  the surrogate for assessment of the painfulness of the procedure
Follow-up-30s | procedure
  absence any arrhythmia recurrence (AR) defined as any documented recurrence of AF and/or atrial tachycardia (AT) and /or atrial flutter (AFL) lasting longer than 30 second

CONTACTS AND LOCATIONS:
Overall Officials: MACIEJ MACIEJ, MD, Principal Investigator — MEDICAL UNIVERSITY OF LUBLIN, POLAND
Locations (1):
- Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D. 2012 HRS/EHRA/ECAS Expert Consensus Statement on Catheter and Surgical Ablation of Atrial Fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design. Europace. 2012 Apr;14(4):528-606. doi: 10.1093/europace/eus027. Epub 2012 Mar 1. No abstract available. PMID 22389422
- [Result] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Alexandru Popescu B, Schotten U, Van Putte B, Vardas P. 2016 ESC Guidelines for the Management of Atrial Fibrillation Developed in Collaboration With EACTS. Rev Esp Cardiol (Engl Ed). 2017 Jan;70(1):50. doi: 10.1016/j.rec.2016.11.033. No abstract available. English, Spanish. PMID 28038729
- [Result] Galeazzi M, Ficili S, Dottori S, Elian MA, Pasceri V, Venditti F, Russo M, Lavalle C, Pandozi A, Pandozi C, Santini M. Pain perception during esophageal warming due to radiofrequency catheter ablation in the left atrium. J Interv Card Electrophysiol. 2010 Mar;27(2):109-15. doi: 10.1007/s10840-009-9447-y. Epub 2009 Nov 27. PMID 19943098
- [Result] Aryana A, Heist EK, D'Avila A, Holmvang G, Chevalier J, Ruskin JN, Mansour MC. Pain and anatomical locations of radiofrequency ablation as predictors of esophageal temperature rise during pulmonary vein isolation. J Cardiovasc Electrophysiol. 2008 Jan;19(1):32-8. doi: 10.1111/j.1540-8167.2007.00975.x. Epub 2007 Sep 24. PMID 17900251
- [Result] Patel PJ, Padanilam BJ. High-power short-duration ablation: Better, safer, and faster? J Cardiovasc Electrophysiol. 2018 Nov;29(11):1576-1577. doi: 10.1111/jce.13749. Epub 2018 Oct 25. No abstract available. PMID 30357991
- [Result] Winkle RA, Mohanty S, Patrawala RA, Mead RH, Kong MH, Engel G, Salcedo J, Trivedi CG, Gianni C, Jais P, Natale A, Day JD. Low complication rates using high power (45-50 W) for short duration for atrial fibrillation ablations. Heart Rhythm. 2019 Feb;16(2):165-169. doi: 10.1016/j.hrthm.2018.11.031. PMID 30712645